CLINICAL TRIAL: NCT06086132
Title: Detection and Prevention of Cancer-Related Cardiovascular Toxicity Registry (ISACS CARDIONCO-PREDICT)
Brief Title: Detection and Prevention of Cancer-Related Cardiovascular Toxicity Registry
Status: Recruiting | Type: Observational
Sponsor: University of Bologna (Other)
Collaborators: Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Responsible Party: Principal Investigator, Olivia Manfrini, MD, Professor, University of Bologna
Other Study IDs: ISACS CARDIONCO-PREDICT
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Cancer Related Cardiovascular Toxicity
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer: Newly diagnosed breast cancer undergoing treatment with anthracyclines analogues with or without radiotherapy, with or without trastuzumab, or other anticancer drugs.
  (Non-interventional prospective patient registry)
  Interventions: Combination Product: Prospective validation of the HFA-ICOS risk score in a subset of subjects with newly diagnosed breast cancer and undergoing treatment with anthracyclines analogues with or without radiotherapy
- Female and Male: Diagnosis of cancer scheduled for treatment according to the treating physician's discretion.
  (Non-interventional patient registry)

INTERVENTIONS:
Combination Product: Prospective validation of the HFA-ICOS risk score in a subset of subjects with newly diagnosed breast cancer and undergoing treatment with anthracyclines analogues with or without radiotherapy — Follow-up visits at baseline, 3-months, and 1-year
  Other Names: Non-interventional patient registry
  Groups: Breast cancer

SUMMARY:
This study is being done in order to assess the cardiovascular events known as cardiovascular toxicity of chemotherapy agents and radiotherapy protocols in cancer subjects to identify risk prediction, prevention and treatment of cancer therapy-related cardiovascular toxicity and cancer therapy-related cardiac dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older
* Capable of giving informed consent
* Diagnosis of cancer scheduled for treatment according to treating physician's discretion
* Life expectancy >1 year
* For the prospective validation of HFA-ICOS risk score validation: Newly diagnosed breast cancer undergoing treatment with anthracyclines analogues with or without radiotherapy, with or without trastuzumab, or other anticancer drugs

Exclusion Criteria:

* Age <18 years old
* Not able to give informed consent
* Life expectancy <1 year
* Advanced-stage cancer not eligible for treatment (subjects with an indication of palliative care) according to treating physician's

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Confirmed diagnosis of cancer undergoing treatment
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
All causes mortality | For approximately a median of 3 years
  Occurrence of all cause death
Cardiovascular mortality | For approximately a median of 3 years
  Occurrence of cardiovascular mortality
Cancer therapy-related cardiovascular toxicity | For approximately a median of 3 years
  Occurrence of cancer therapy-related cardiovascular toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Olivia Manfrini, MD, Principal Investigator — University of Bologna; Prof. Giuseppina Novo, MD, Principal Investigator — Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone
Locations (5):
- Italy (2):
  - University of Bologna, Bologna
  - Azienda Ospedaliera Universitaria Policlinico "Paolo Giaccone", Palermo
- Ss. Cyril and Methodius University in Skopje, University Clinic, Skopje, North Macedonia
- Serbia (2):
  - University of Belgrade, Clinical Center of Serbia, Belgrade
  - University of Belgrade, Clinical Hospital Center Bezanijska kosa, Belgrade

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lyon AR, Lopez-Fernandez T, Couch LS, Asteggiano R, Aznar MC, Bergler-Klein J, Boriani G, Cardinale D, Cordoba R, Cosyns B, Cutter DJ, de Azambuja E, de Boer RA, Dent SF, Farmakis D, Gevaert SA, Gorog DA, Herrmann J, Lenihan D, Moslehi J, Moura B, Salinger SS, Stephens R, Suter TM, Szmit S, Tamargo J, Thavendiranathan P, Tocchetti CG, van der Meer P, van der Pal HJH; ESC Scientific Document Group. 2022 ESC Guidelines on cardio-oncology developed in collaboration with the European Hematology Association (EHA), the European Society for Therapeutic Radiology and Oncology (ESTRO) and the International Cardio-Oncology Society (IC-OS). Eur Heart J. 2022 Nov 1;43(41):4229-4361. doi: 10.1093/eurheartj/ehac244. No abstract available. PMID 36017568